CLINICAL TRIAL: NCT03431350
Title: A Phase 1b-2 Study of Niraparib Combination Therapies for the Treatment of Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of Niraparib Combination Therapies for the Treatment of Metastatic Castration-Resistant Prostate Cancer
Acronym: QUEST
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108406; 64091742PCR2002 (Other: Janssen Research & Development, LLC); 2017-003552-23 (EudraCT Number)
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — niraparib; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Combination 1:Dose Selection: Niraparib + cetrelimab (Part 1) (Experimental): Dose regimen 1: The participants will receive niraparib 200 milligram (mg) orally once daily in combination with cetrelimab 240 mg intravenously (IV) once every 2 weeks. Dose regimen 2: The participants will receive niraparib 200 mg orally once daily in combination with cetrelimab 480 mg IV once every 4 weeks in 28-day treatment cycles until disease progression, unacceptable toxicity, death, or the sponsor terminates the study. The safety evaluation team (SET) will determine if an additional cohort is necessary, based on the data from dose regimens 1 and 2. Participants in the Treatment Phase of this combination will be offered the option to enter the Long-term Extension Phase of the study.
  Interventions: Drug: Niraparib 200 mg; Drug: Cetrelimab 240 mg; Drug: Cetrelimab 480 mg
- Combination 1:Dose Expansion: Niraparib + cetrelimab (Part 2) (Experimental): Participants will be assigned to either Cohort 1A (Biomarker [BM] positive [+]) or Cohort 1B (BM negative [-]) and will receive established RP2D of cetrelimab and niraparib, in Part 2 until disease progression, unacceptable toxicity, death, or the sponsor terminates the study. A futility analysis will be performed for the Cohort 1B after 10 BM- participants are enrolled in Part 2. This cohort will be closed if the response is less than predetermined response rate as outlined in the protocol. Participants in the Treatment Phase of this combination will be offered the option to enter the Long-term Extension Phase of the study.
  Interventions: Drug: Niraparib 200 mg; Drug: Cetrelimab 480 mg
- Combination 2: Dose Expansion: Niraparib + AA-P (Part 2) (Experimental): Participants will be assigned to one of 4 cohorts based on biomarker status - Cohort 2A (BRCA biallelic loss), 2B (other DRD biallelic loss), 2C (BRCA monoallelic loss), or 2D (other DRD monoallelic loss), and will receive niraparib 200 mg once daily in combination with abiraterone acetate 1000 mg (4*250 mg) plus 10 mg prednisone (5 mg twice daily) throughout treatment phase. Participants in the Treatment Phase of this combination will be offered the option to enter the Long-term Extension Phase of the study.
  Interventions: Drug: Niraparib 200 mg; Drug: Abiraterone acetate 1000 mg; Drug: Prednisone 5 mg
- Combination 3: Niraparib + AA-P (Experimental): Participants will be assigned to one of three cohorts to receive AA-P with or without niraparib. Participants in the Treatment Phase of this combination will be offered the option to enter the Long-term Extension Phase of the study.
  Interventions: Drug: Niraparib 200 mg; Drug: Abiraterone acetate 1000 mg; Drug: Prednisone 5 mg

INTERVENTIONS:
Drug: Niraparib 200 mg — Participants will receive niraparib 200 mg orally.
Drug: Cetrelimab 240 mg — Participants will receive cetrelimab 240 mg IV every 2 weeks.
  Other Names: JNJ-63723283
  Arms: Combination 1:Dose Selection: Niraparib + cetrelimab (Part 1)
Drug: Cetrelimab 480 mg — Participants will receive cetrelimab 480 mg IV every 4 weeks.
  Other Names: JNJ-63723283
  Arms: Combination 1:Dose Expansion: Niraparib + cetrelimab (Part 2); Combination 1:Dose Selection: Niraparib + cetrelimab (Part 1)
Drug: Abiraterone acetate 1000 mg — Participants will receive AA 1000 mg orally.
  Arms: Combination 2: Dose Expansion: Niraparib + AA-P (Part 2); Combination 3: Niraparib + AA-P
Drug: Prednisone 5 mg — Participants will receive prednisone 5 mg orally.
  Arms: Combination 2: Dose Expansion: Niraparib + AA-P (Part 2); Combination 3: Niraparib + AA-P

SUMMARY:
The purpose of this study is to: a) establish the recommended phase 2 dose (RP2D) and to evaluate the antitumor activity and safety of niraparib combination therapies (Combinations 1 and 2) and b) to determine the relative bioavailability of niraparib and abiraterone acetate (AA) in combination (Combination 3) in participants with metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This multicenter study will evaluate safety and efficacy of niraparib in combination with other anti-cancer agents. Combination 1 will combine niraparib with the anti-programmed cell death protein (PD)-1 monoclonal antibody cetrelimab, in participants with mCRPC. Combination 1 has 2 parts: in Part 1 (dose selection), participants will be enrolled to establish RP2D doses of niraparib and cetrelimab; and Part 2 (dose expansion) will evaluate the combination therapy in an expanded number of participants into 2 cohorts (biomarker positive or biomarker negative). Combination 2 will combine niraparib with abiraterone acetate plus prednisone (AA-P) in mCRPC participants with DNA-repair gene defects (DRD). Combination 3 will evaluate the relative bioavailability (BA) of niraparib and AA in combination. In a pharmacokinetics (PK) assessment phase, niraparib and AA will be administered, and in an extension phase, niraparib and AA-P will be administered. Combinations 1 and 2 will have 5 phases: A Pre-screening Phase, a Screening Phase, a Treatment Phase, a Follow-up Phase, and a Long-term Extension (LTE) Phase; Combination 3 has 3 phases: A Screening Phase, A PK Assessment Phase, an Extension Phase (including LTE phase). Study evaluations will include efficacy, PK, PK/pharmacodynamics, biomarkers, safety and tolerability.

ELIGIBILITY:
Inclusion Criteria for Combination 3:

* Diagnosed with mCRPC, who in the opinion of the investigator may benefit from treatment in Combination 3 of this study
* Able to continue gonadotropin releasing hormone analogue (GnRHa) therapy during the study if not surgically castrate (that is, subjects who has not undergone bilateral orchiectomy).
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of less than or equal to (<=) 1
* Toxicity associated with prior chemotherapy or radiotherapy has resolved to Grade <= 1 (except alopecia or Grade <= 2 neuropathy) at screening
* Participant must agree not to donate sperm while on study treatment, and for 3 months following the last dose of study treatment

Exclusion Criteria:

* History or current diagnosis of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML)
* Active malignancies (that is, progressing or requiring treatment change in the last 24 months) other than the disease being treated under study. The only allowed exceptions are: non-muscle invasive bladder cancer; skin cancer (non-melanoma or melanoma); breast cancer; malignancy that is considered cured with minimal risk of recurrence
* Active infection requiring systemic therapy
* Allergies, hypersensitivity, or intolerance to niraparib or the corresponding excipients

Combination 3:

* Symptomatic brain metastases
* Prior disease progression during combination treatment with AA and poly (adenosine diphosphate [ADP]-ribose) polymerase inhibitor (PARPi). Prior discontinuation of treatment with AA or PARPi due to AA- or PARPi-related toxicity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (50):
- United States (19):
  - Urological Associates of Southern Arizona, P.C., Tucson, Arizona
  - The Urology Center of Colorado, Denver, Colorado
  - Mayo Clinic - Division Of Hematology/oncology, Jacksonville, Florida
  - First Urology, PSC, Jeffersonville, Indiana
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Michigan Institute of Urology, Troy, Michigan
  - New York Oncology Hematology, Albany, New York
  - Memorial Sloan Kettering Cancer Center, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - MUSC-Hollings Cancer Center, Charleston, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, Nashville, Tennessee
  - Houston Metro Urology, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Urology of Virginia, PLCC, Virginia Beach, Virginia
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Belgium (6):
  - OLV Ziekenhuis Aalst, Aalst
  - ZNA Middelheim, Antwerp
  - ULB Hôpital Erasme, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Az Groeninge, Kortrijk
  - Centre Hospitalier Universitaire de Liege Domaine Universitaire du Sart Tilman, Liège
- Canada (4):
  - Southern Alberta Institute of Urology / Prostate Cancer Centre, Calgary, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Princess Margaret Cancer Centre University Health Network, Toronto, Ontario
  - Centre de Recherche du CHUM, Montreal, Quebec
- Israel (5):
  - Asaf Harofe Medical Center, Beer Yaakov
  - Soroka Hospital, Beersheba
  - Rambam Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center Tel Hashomer, Ramat Gan
- Italy (5):
  - Azienda Ospedaliera Universitaria Careggi di Firenze, Florence
  - Azienda Ospedaliera ''Vito Fazzi'', Lecce
  - UOC Oncologia Ospedale Provinciale di Macerata, Macerata
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - IRCCS-Fondazione Pascale, Napoli
- Spain (6):
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hospital Vall D'Hebron, Barcelona
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid
  - Hosp Virgen de La Victoria, Málaga
- United Kingdom (5):
  - Royal United Hospital, Bath
  - University College London Hospitals, London
  - Southampton General Hospital, Southampton
  - The Royal Marsden NHS Trust Sutton, Sutton
  - Royal Cornwall Hospitals NHS Trust - Royal Cornwall Hospital, Truro

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Combination 2, one participant who was homologous recombination repair (HRR) negative was erroneously enrolled to Cohort 2C (BRCA monoallelic loss) and thus was not included in the Intent-to-Treat (ITT) Population for the efficacy analysis. but was included in the safety analysis. This participant data were presented in participant flow, baseline characteristics and adverse events section. Data reported based on primary completion date, i.e., August 31, 2021.
Groups:
- Combination 1: Part 1 (Dose Seletion): Niraparib 200 mg + Cetrelimab 240 mg: Participants with metastatic castration-resistant prostate cancer (mCRPC) who were either biomarker positive (BM+) or BM negative (BM-) for deoxyribonucleic acid (DNA)-repair gene defects (DRD) or BM+ for cyclin-dependent kinase 12 (CDK12) pathogenic alterations received niraparib 200 milligrams (mg) orally once daily in combination with cetrelimab 240 mg intravenous (IV) once every 4 weeks (i.e., on Day 1 of each cycle) in each 28-day treatment cycle until disease progression, unacceptable toxicity, death, or the sponsor terminated the study.
- Combination 1: Part 1 (Dose Selection): Niraparib 200 mg + Cetrelimab 480 mg: Participants with mCRPC who were either BM+ or BM- for DRD or BM+ for CDK12 pathogenic alterations received niraparib 200 mg orally once daily in combination with cetrelimab 480 mg IV infusion once every 4 weeks (i.e., on Day 1 of each cycle) in each 28-day treatment cycle until disease progression, unacceptable toxicity, death, or the sponsor terminated the study.
- Combination 1: Part 2 (Dose Expansion): Cohort 1A: BM+: Niraparib 200 mg + Cetrelimab 480 mg: Participants with mCRPC and were BM+ received established recommended Phase 2 dose (RP2D) of niraparib 200 mg once daily in combination with cetrelimab 480 mg IV infusion every 4 weeks i.e., on Day 1 of each cycle) in each 28-day treatment cycle until disease progression, unacceptable toxicity, death, or the sponsor terminated the study.
- Combination 1: Part 2 (Dose Expansion): Cohort 1B: BM-: Niraparib 200 mg + Cetrelimab 480 mg: Participants with mCRPC and were BM- received established RP2D of niraparib 200 mg once daily in combination with cetrelimab 480 mg IV infusion every 4 weeks i.e., on Day 1 of each cycle) in each 28-day treatment cycle until disease progression, unacceptable toxicity, death, or the sponsor terminated the study.
- Combination 2: Cohort 2A: Niraparib+Abiraterone Acetate+Prednisone: Participants with mCRPC and HRR gene alterations (breast cancer gene [BRCA] biallelic loss [2A]) received niraparib 200 mg orally once daily in combination with abiraterone acetate 1000 mg orally once daily plus prednisone (P) 10 mg (2*5 mg) orally twice daily in each 28-day treatment cycle until disease progression, unacceptable toxicity, death, or the sponsor terminated the study.
- Combination 2: Cohort 2C: Niraparib+Abiraterone Acetate+Prednisone: Participants with mCRPC and HRR gene alterations (BRCA monoallelic loss [2C]) received niraparib 200 mg orally once daily in combination with abiraterone acetate 1000 mg orally once daily plus prednisone 10 mg (2*5 mg) orally twice daily in each 28-day treatment cycle until disease progression, unacceptable toxicity, death, or the sponsor terminated the study.
- Combination 2: Cohort 2D: Niraparib+Abiraterone Acetate+Prednisone: Participants with mCRPC and HRR gene alterations (other DRD monoallelic loss [2D]) received niraparib 200 mg orally once daily in combination with abiraterone acetate 1000 mg orally once daily plus prednisone 10 mg (2*5 mg) orally twice daily in each 28-day treatment cycle until disease progression, unacceptable toxicity, death, or the sponsor terminated the study.
- Combination 2: Cohort 2C: HRR Negative: Niraparib + Abiraterone Acetate + Prednisone: Participants with mCRPC and HRR gene alteration negative received niraparib 200 mg orally once daily in combination with abiraterone acetate 1000 mg orally once daily plus prednisone 10 mg (2*5 mg) orally twice daily in each 28-day treatment cycle until disease progression, unacceptable toxicity, death, or the sponsor terminated the study.
- Combination 3: Cohort 1A: Niraparib + Abiraterone Acetate, SA: Participants with mCRPC (regardless of HRR BM status) received a single dose of niraparib 200 mg in combination with single oral dose of abiraterone acetate 1000 mg as single agent (SA) orally from Cycle 1 Day 1 to Day 8. After completion of Cycle 1 Day 8 (Pharmacokinetic [PK] Assessment Phase), Participants had the option to enter the Long-term Extension Phase of the study and received protocol defined treatment until study discontinuation.
- Combination 3: Cohort 1B: Niraparib + Abiraterone Acetate, FDC1-RS (G010): Participants with mCRPC received a single dose of niraparib 200 mg in combination with single oral dose of abiraterone acetate 1000 as fixed-dose combination 1 (FDC1) regular-strength (RS) tablets orally from Cycle 2 1 Day 1 to Day 8. After completion of Cycle 1 Day 8 (PK Assessment Phase), participants had an option to enter the Long-term Extension Phase of the study and received protocol defined treatment until study discontinuation.
- Combination 3: Cohort 2: Niraparib + Abiraterone Acetate, FDC2-RS (G012): Participants with mCRPC received a single dose of niraparib 200 mg in combination with single oral dose of abiraterone acetate 1000 mg as FDC2 RS tablets orally from Cycle 2 1 Day 1 to Day 8. After completion of Cycle 1 Day 8 (PK Assessment Phase), participants had an option to enter the Long-term Extension Phase of the study and received protocol defined treatment until study discontinuation.
- Combination 3: Cohort 3: Niraparib + Abiraterone Acetate, FDC1-LS: Participants with mCRPC received a single oral dose of niraparib 100 mg in combination with single oral dose of abiraterone acetate 1000 mg as FDC1 low strength (LS) tablets orally from Cycle 2 1 Day 1 to Day 8. After completion of Cycle 1 Day 8 (PK Assessment Phase), participants had an option to enter the Long-term Extension Phase of the study and received protocol defined treatment until study discontinuation.
Period: Overall Study
Arm/Group | Combination 1: Part 1 (Dose Seletion): Niraparib 200 mg + Cetrelimab 240 mg | Combination 1: Part 1 (Dose Selection): Niraparib 200 mg + Cetrelimab 480 mg | Combination 1: Part 2 (Dose Expansion): Cohort 1A: BM+: Niraparib 200 mg + Cetrelimab 480 mg | Combination 1: Part 2 (Dose Expansion): Cohort 1B: BM-: Niraparib 200 mg + Cetrelimab 480 mg | Combination 2: Cohort 2A: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2C: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2D: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2C: HRR Negative: Niraparib + Abiraterone Acetate + Prednisone | Combination 3: Cohort 1A: Niraparib + Abiraterone Acetate, SA | Combination 3: Cohort 1B: Niraparib + Abiraterone Acetate, FDC1-RS (G010) | Combination 3: Cohort 2: Niraparib + Abiraterone Acetate, FDC2-RS (G012) | Combination 3: Cohort 3: Niraparib + Abiraterone Acetate, FDC1-LS
Started | 6 | 6 | 21 | 11 | 8 | 9 | 6 | 1 | 17 | 17 | 17 | 17
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 21 | 11 | 8 | 9 | 6 | 1 | 17 | 17 | 17 | 17
Not completed — ONGOING | 0 | 0 | 2 | 0 | 1 | 3 | 0 | 1 | 3 | 4 | 2 | 1
Not completed — Death | 6 | 5 | 18 | 7 | 4 | 3 | 2 | 0 | 0 | 0 | 4 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Other | 0 | 0 | 1 | 3 | 2 | 2 | 4 | 0 | 14 | 11 | 11 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination 1: Part 1 (Dose Seletion): Niraparib 200 mg + Cetrelimab 240 mg | Combination 1: Part 1 (Dose Selection): Niraparib 200 mg + Cetrelimab 480 mg | Combination 1: Part 2 (Dose Expansion): Cohort 1A: BM+: Niraparib 200 mg + Cetrelimab 480 mg | Combination 1: Part 2 (Dose Expansion): Cohort 1B: BM-: Niraparib 200 mg + Cetrelimab 480 mg | Combination 2: Cohort 2A: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2C: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2D: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2C: HRR Negative: Niraparib + Abiraterone Acetate + Prednisone | Combination 3: Cohort 1A: Niraparib + Abiraterone Acetate, SA | Combination 3: Cohort 1B: Niraparib + Abiraterone Acetate, FDC1-RS (G010) | Combination 3: Cohort 2: Niraparib + Abiraterone Acetate, FDC2-RS (G012) | Combination 3: Cohort 3: Niraparib + Abiraterone Acetate, FDC1-LS | Total
Number analyzed (Participants) | 6 | 6 | 21 | 11 | 8 | 9 | 6 | 1 | 17 | 17 | 17 | 17 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (7.15) | 66.7 (12.56) | 68.1 (6.6) | 66.6 (3.91) | 71.4 (8.23) | 71.3 (5.89) | 72.8 (9.75) | 80 | 72.3 (7.19) | 71.1 (7.96) | 71.2 (7.85) | 72.9 (7.36) | 70.4 (7.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 21 | 11 | 8 | 9 | 6 | 1 | 17 | 17 | 17 | 17 | 136
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Black or African American | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 5 | 6 | 21 | 8 | 7 | 9 | 5 | 0 | 14 | 14 | 16 | 16 | 121
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 4 | 2 | 4 | 3 | 16
  CANADA | 0 | 0 | 3 | 0 | 1 | 4 | 2 | 0 | 2 | 2 | 2 | 0 | 16
  ISRAEL | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 7 | 5 | 2 | 8 | 27
  ITALY | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  SPAIN | 2 | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 13
  UNITED KINGDOM | 3 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 8
  UNITED STATES | 1 | 2 | 8 | 8 | 4 | 4 | 3 | 1 | 4 | 8 | 4 | 6 | 53

OUTCOME MEASURES:

1. Primary Outcome: Combination 1: Part 1: Number of Participants With Specified Toxicity
Description: Number of participants with specified toxicity during Cycle 1 was reported. Only toxicities that occurred during safety evaluation period(defined as first 28 days of treatment-Cycle 1 of Part 1) was used for analysis of specified toxicities and for dose reduction decisions. Toxicities were graded for severity as per NCI-CTCAE, version 4.03. Safety evaluation criteria were: Any Grade(G) >=3 non-hematological toxicity without anorexia, or constipation, fatigue improved to G<=2 in <7 days, vomiting and diarrhea resolved in <=3 days, laboratory abnormalities with hospitalization, tumor flare improved to G<=2 in <=7 days, elevation in AST/ALT for <=7 days and G3 hypertension controlled by medical therapy; any treatment-related(TR)G4 or G>=3 thrombocytopenia required platelet transfusion; Any TR G4 neutropenia >=7 days or G3 or 4 neutropenia with infection/fever >38.5 degrees Celsius; Any TR SAE or intolerable toxicity.
Time Frame: Cycle 1 (28 days)
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure. This outcome measure was analyzed for specified arms only as pre-planned in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination 1: Part 1 (Dose Seletion): Niraparib 200 mg + Cetrelimab 240 mg | Combination 1: Part 1 (Dose Selection): Niraparib 200 mg + Cetrelimab 480 mg
Number analyzed (Participants) | 5 | 6
Participants | 0 | 0

2. Primary Outcome: Combination 1: Part 2: Objective Response Rate (ORR)
Description: ORR of soft tissue (visceral or nodal disease) was defined as percentage of participants with measurable disease who achieved a best response of either complete response (CR) or partial response (PR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 with no evidence of bone progression according to prostate cancer working group 3 (PCWG3) criteria.
Time Frame: Up to 37 months
Population: Intent-to-Treat (ITT) analysis set included all participants who had at least 1 dose of both study drugs at the selected RP2D in Combination 1: Part 2 of study. This outcome measure was analyzed for specified arms only as pre-planned in the protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combination 1: Part 2 (Dose Expansion): Cohort 1A: BM+: Niraparib 200 mg + Cetrelimab 480 mg | Combination 1: Part 2 (Dose Expansion): Cohort 1B: BM-: Niraparib 200 mg + Cetrelimab 480 mg
Number analyzed (Participants) | 21 | 11
Percentage of participants | 23.8 [9.9 to 43.7] | 9.1 [0.5 to 36.4]

3. Primary Outcome: Combination 2: Composite Response Rate (RR)
Description: Composite response rate was defined as the percentage of participants who had a composite response which is defined as one of the following PCWG3 criteria: Objective response (percentage of participants with measurable disease who achieved a best response of either CR or PR as assessed by RECIST 1.1 with no evidence of bone progression according to PCWG3 criteria) (confirmed per RECIST 1.1), or; circulating tumor cells (CTC) response: defined as CTC=0 per 7.5 milliliters (mL) of blood at 8 weeks for participants who had CTC greater than or equal to (>=) 1 at baseline or CTC less than (<) 5 per 7.5 mL with CTC >=5 at baseline, confirmed by a second consecutive value obtained 4 or more weeks later, or prostate-specific antigen (PSA) declined of >=50 percentage (%), measured twice 3 to 4 weeks apart. This outcome measure was analyzed for specified arms only as pre-planned in the protocol.
Time Frame: Up to 31 months
Population: ITT analysis set included all participants who had at least 1 dose of both study drugs at the selected RP2D in Part 2 of study. In Combination 2, one participant who was HRR negative was erroneously enrolled to Cohort 2C (BRCA monoallelic loss) and was presented under arm named "Combination 2: Cohort 2C: HRR negative: Niraparib + Abiraterone Acetate + Prednisone". Due to erroneous enrollment, this participant was not included in the ITT population for the efficacy analysis of this endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combination 2: Cohort 2A: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2C: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2D: Niraparib+Abiraterone Acetate+Prednisone
Number analyzed (Participants) | 8 | 9 | 6
Percentage of participants | 75.0 [40.0 to 95.4] | 55.6 [25.1 to 83.1] | 33.3 [6.3 to 72.9]

4. Primary Outcome: Combination 1: Part 2: Number of Participants With Adverse Events (AEs)
Description: AE was defined as an any untoward medical occurrence in a clinical study subject administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment.
Time Frame: Up to 37 months
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug. This outcome measure was analyzed for specified arms only as pre-planned in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination 1: Part 2 (Dose Expansion): Cohort 1A: BM+: Niraparib 200 mg + Cetrelimab 480 mg | Combination 1: Part 2 (Dose Expansion): Cohort 1B: BM-: Niraparib 200 mg + Cetrelimab 480 mg
Number analyzed (Participants) | 21 | 11
Participants | 21 | 11

5. Primary Outcome: Combination 2: Number of Participants With Adverse Events (AEs)
Description: as for outcome 4
Time Frame: Up to 31 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Combination 2: Cohort 2A: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2C: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2D: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2C: HRR Negative: Niraparib + Abiraterone Acetate + Prednisone
Number analyzed (Participants) | 8 | 9 | 6 | 1
Participants | 8 | 9 | 5 | 1

6. Primary Outcome: Combination 1: Part 2: Number of Participants With Adverse Events (AEs) of Grade >=3 Severity
Description: AE was defined as an any untoward medical occurrence in a clinical study subject administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An assessment of severity grade was made using the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) as Grade 1 (mild): awareness of symptoms that are easily tolerated, causing minimal discomfort and not interfering with everyday activities; Grade 2 (moderate): sufficient discomfort is present to cause interference with normal activity; Grade 3 (severe): extreme distress, causing significant impairment of functioning or incapacitation, prevents normal everyday activities; Grade 4 (Life-threatening): urgent intervention indicated; and Grade 5 (death).
Time Frame: Up to 37 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Combination 1: Part 2 (Dose Expansion): Cohort 1A: BM+: Niraparib 200 mg + Cetrelimab 480 mg | Combination 1: Part 2 (Dose Expansion): Cohort 1B: BM-: Niraparib 200 mg + Cetrelimab 480 mg
Number analyzed (Participants) | 21 | 11
Participants | 14 | 8

7. Primary Outcome: Combination 2: Number of Participants With Adverse Events (AEs) of Grade >=3 Severity
Description: AE was defined as an any untoward medical occurrence in a clinical study subject administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An assessment of severity grade was made using the NCI-CTCAE as Grade 1 (mild): awareness of symptoms that are easily tolerated, causing minimal discomfort and not interfering with everyday activities; Grade 2 (moderate): sufficient discomfort is present to cause interference with normal activity; Grade 3 (severe): extreme distress, causing significant impairment of functioning or incapacitation, prevents normal everyday activities; Grade 4 (Life-threatening): urgent intervention indicated; and Grade 5 (death).
Time Frame: Up to 31 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Combination 2: Cohort 2A: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2C: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2D: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2C: HRR Negative: Niraparib + Abiraterone Acetate + Prednisone
Number analyzed (Participants) | 8 | 9 | 6 | 1
Participants | 6 | 7 | 4 | 1

8. Primary Outcome: Combination 3: Maximum Observed Plasma Concentration (Cmax) of Niraparib and Abiraterone Acetate After a Single Dose
Description: Cmax is defined as maximum observed plasma concentration of niraparib and abiraterone acetate (AA) after a single dose.
Time Frame: Pre-dose, 30 min, 1 hour (hr), 1.5 hr, 2hr, 3 hr, 4 hr, 6 hr, 8 hr, 10 hr, 24 hr, 48 hr, 72 hr, and 168 hr post dose on Day 1
Population: Pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of both study agents (either as a fixed dose combination [FDC] or single agent combination [SAC]) and had at least 1 concentration value. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure. This outcome measure was analyzed for specified arms only as pre-planned in the protocol.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Combination 3: Cohort 1A: Niraparib + Abiraterone Acetate, SA | Combination 3: Cohort 1B: Niraparib + Abiraterone Acetate, FDC1-RS (G010) | Combination 3: Cohort 2: Niraparib + Abiraterone Acetate, FDC2-RS (G012)
Number analyzed (Participants) | 16 | 16 | 17
Nanograms per milliliter (ng/mL) | 428 (189) | 398 (160) | 417 (176)

9. Primary Outcome: Combination 3: Maximum Observed Plasma Concentration (Cmax) of Niraparib Normalized by the Dose(Niraparib) (Cmax/Dose) of Niraparib Administered With AA After a Single Dose
Description: Cmax/dose of niraparib was defined as maximum observed plasma concentration of niraparib Cmax normalized by the dose of niraparib administered with AA after a single dose.
Time Frame: as for outcome 8
Population: PK analysis set included all participants who received at least 1 dose of both study agents (either as a FDC or SAC) and had at least 1 concentration value. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure. This outcome measure was analyzed for specified arms only as pre-planned in the protocol.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter per milligram
Arm/Group | Combination 3: Cohort 1A: Niraparib + Abiraterone Acetate, SA | Combination 3: Cohort 1B: Niraparib + Abiraterone Acetate, FDC1-RS (G010) | Combination 3: Cohort 2: Niraparib + Abiraterone Acetate, FDC2-RS (G012)
Number analyzed (Participants) | 16 | 16 | 17
nanograms per milliliter per milligram | 2.14 (0.95) | 1.99 (0.80) | 2.09 (0.88)

10. Primary Outcome: Combination 3: Area Under the Plasma Concentration-Time Curve From Time Zero to 168 Hours (AUC [0-168hr]) of Niraparib Administered With AA After a Single Dose
Description: AUC(0-168 hours) was defined as area under the plasma concentration-time curve from time zero to 168 hours of Niraparib administered with AA After a single dose.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Nanograms*hour per milliliter (ng*h/mL)
Arm/Group | Combination 3: Cohort 1A: Niraparib + Abiraterone Acetate, SA | Combination 3: Cohort 1B: Niraparib + Abiraterone Acetate, FDC1-RS (G010) | Combination 3: Cohort 2: Niraparib + Abiraterone Acetate, FDC2-RS (G012)
Number analyzed (Participants) | 16 | 15 | 17
Nanograms*hour per milliliter (ng*h/mL) | 14672 (7346) | 11862 (4973) | 13321 (5843)

11. Primary Outcome: Combination 3: Area Under the Plasma Concentration-Time Curve for Niraparib From Time Zero to 168 Hours (AUC [0-168 Hours]/Dose) of Niraparib Administered With AA After a Single Dose
Description: AUC0(168 hours)/dose was defined as area under the plasma concentration-time curve for niraparib from time 0 to 168 hours of niraparib administered with AA after a single dose.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter/milligram
Arm/Group | Combination 3: Cohort 1A: Niraparib + Abiraterone Acetate, SA | Combination 3: Cohort 1B: Niraparib + Abiraterone Acetate, FDC1-RS (G010) | Combination 3: Cohort 2: Niraparib + Abiraterone Acetate, FDC2-RS (G012)
Number analyzed (Participants) | 16 | 16 | 17
nanogram*hour/milliliter/milligram | 73.36 (36.73) | 59.31 (24.87) | 66.61 (29.22)

12. Secondary Outcome: Combination 1: Parts 1 and 2: Plasma Concentrations of Niraparib
Time Frame: Day 1
Reporting Status: Not Posted, anticipated posting 2026-12

13. Secondary Outcome: Combination 1: Parts 1 and 2: Maximum Observed Plasma Concentration (Cmax) of Niraparib
Time Frame: Day 1
Reporting Status: Not Posted, anticipated posting 2026-12

14. Secondary Outcome: Combination 1: Parts 1 and 2: Time to Reach the Maximum Plasma Concentration (Tmax) of Niraparib
Time Frame: Day 1
Reporting Status: Not Posted, anticipated posting 2026-12

15. Secondary Outcome: Combination 1: Parts 1 and 2: Minimum Observed (Predose) Concentration Following Multiple Dosing (Ctrough) of Niraparib
Time Frame: Day 1
Reporting Status: Not Posted, anticipated posting 2026-12

16. Secondary Outcome: Combination 1: Parts 1 and 2: Number of Participants With Anti-drug Antibodies of Niraparib
Time Frame: From baseline up to end of study (6 years 10 months)
Reporting Status: Not Posted, anticipated posting 2026-12

17. Secondary Outcome: Combination 1: Part 2 and Combination 2: Circulating Tumor Cells (CTC) Response
Time Frame: From baseline up to end of study (6 years 10 months)
Reporting Status: Not Posted, anticipated posting 2026-12

18. Secondary Outcome: Combination 1: Part 2: Composite Response Rate
Time Frame: From baseline up to end of study (6 years 10 months)
Reporting Status: Not Posted, anticipated posting 2026-12

19. Secondary Outcome: Combination 2: Objective Response Rate (ORR)
Time Frame: From baseline up to end of study (6 years 10 months)
Reporting Status: Not Posted, anticipated posting 2026-12

20. Secondary Outcome: Combination 1: Part 2 and Combination 2: Duration of Objective Response
Time Frame: From baseline up to end of study (6 years 10 months)
Reporting Status: Not Posted, anticipated posting 2026-12

21. Secondary Outcome: Combination 1: Part 2 and Combination 2: Overall Survival
Time Frame: From baseline up to end of study (6 years 10 months)
Reporting Status: Not Posted, anticipated posting 2026-12

22. Secondary Outcome: Combination 3: Cmax of Niraparib and Abiraterone Acetate After a Single Dose For Low-strength FDC
Time Frame: as for outcome 8
Reporting Status: Not Posted, anticipated posting 2026-12

23. Secondary Outcome: Combination 3: Maximum Observed Plasma Concentration (Cmax) of Niraparib Normalized by the Dose(Niraparib) (Cmax/Dose) of Niraparib Administered With AA After a Single Dose for Low-strength FDC
Time Frame: as for outcome 8
Reporting Status: Not Posted, anticipated posting 2026-12

24. Secondary Outcome: Combination 3: Area Under the Plasma Concentration-Time Curve From Time Zero to 168 Hours (AUC [0-168hr]) of Niraparib Administered With AA After a Single Dose For Low-strength FDC
Time Frame: as for outcome 8
Reporting Status: Not Posted, anticipated posting 2026-12

25. Secondary Outcome: Combination 3: Area Under the Plasma Concentration-Time Curve for Niraparib From Time Zero to 168 Hours (AUC [0-168 Hours]/Dose) of Niraparib Administered With AA After a Single Dose For Low-strength FDC
Time Frame: as for outcome 8
Reporting Status: Not Posted, anticipated posting 2026-12

26. Secondary Outcome: Combination 3: Number of Participants With Adverse Events
Time Frame: From baseline up to end of study (6 years 10 months)
Reporting Status: Not Posted, anticipated posting 2026-12

27. Secondary Outcome: Combination 3: Number of Participants With Clinical Laboratory Parameters
Time Frame: From baseline up to end of study (6 years 10 months)
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: Combination 1: Part 1: Up to 42 months and Part 2: up to 37 months; Combination 2: up to 31 months; Combination 3: up to 18 months
Description: The safety analysis set included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Combination 1: Part 1 (Dose Seletion): Niraparib 200 mg + Cetrelimab 240 mg | Combination 1: Part 1 (Dose Selection): Niraparib 200 mg + Cetrelimab 480 mg | Combination 1: Part 2 (Dose Expansion): Cohort 1A: BM+: Niraparib 200 mg + Cetrelimab 480 mg | Combination 1: Part 2 (Dose Expansion): Cohort 1B: BM-: Niraparib 200 mg + Cetrelimab 480 mg | Combination 2: Cohort 2A: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2C: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2D: Niraparib+Abiraterone Acetate+Prednisone | Combination 2: Cohort 2C: HRR Negative: Niraparib + Abiraterone Acetate + Prednisone | Combination 3: Cohort 1A: Niraparib + Abiraterone Acetate, SA | Combination 3: Cohort 1B: Niraparib + Abiraterone Acetate, FDC1-RS (G010) | Combination 3: Cohort 2: Niraparib + Abiraterone Acetate, FDC2-RS (G012) | Combination 3: Cohort 3: Niraparib + Abiraterone Acetate, FDC1-LS
All-Cause Mortality (participants affected / at risk) | 6/6 | 5/6 | 18/21 | 7/11 | 5/8 | 4/9 | 2/6 | 0/1 | 3/17 | 1/17 | 4/17 | 2/17
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/6 | 12/21 | 6/11 | 4/8 | 5/9 | 1/6 | 1/1 | 4/17 | 4/17 | 7/17 | 3/17
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 21/21 | 11/11 | 8/8 | 9/9 | 5/6 | 1/1 | 10/17 | 10/17 | 6/17 | 5/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination 1: Part 1 (Dose Seletion): Niraparib 200 mg + Cetrelimab 240 mg (N=6) | Combination 1: Part 1 (Dose Selection): Niraparib 200 mg + Cetrelimab 480 mg (N=6) | Combination 1: Part 2 (Dose Expansion): Cohort 1A: BM+: Niraparib 200 mg + Cetrelimab 480 mg (N=21) | Combination 1: Part 2 (Dose Expansion): Cohort 1B: BM-: Niraparib 200 mg + Cetrelimab 480 mg (N=11) | Combination 2: Cohort 2A: Niraparib+Abiraterone Acetate+Prednisone (N=8) | Combination 2: Cohort 2C: Niraparib+Abiraterone Acetate+Prednisone (N=9) | Combination 2: Cohort 2D: Niraparib+Abiraterone Acetate+Prednisone (N=6) | Combination 2: Cohort 2C: HRR Negative: Niraparib + Abiraterone Acetate + Prednisone (N=1) | Combination 3: Cohort 1A: Niraparib + Abiraterone Acetate, SA (N=17) | Combination 3: Cohort 1B: Niraparib + Abiraterone Acetate, FDC1-RS (G010) (N=17) | Combination 3: Cohort 2: Niraparib + Abiraterone Acetate, FDC2-RS (G012) (N=17) | Combination 3: Cohort 3: Niraparib + Abiraterone Acetate, FDC1-LS (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 2 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
General Physical Health Deterioration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corona Virus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Enterocolitis Infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes Simplex Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyonephrosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour Compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral Ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device Dislocation (Product Issues) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device Occlusion (Product Issues) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic Venous Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination 1: Part 1 (Dose Seletion): Niraparib 200 mg + Cetrelimab 240 mg (N=6) | Combination 1: Part 1 (Dose Selection): Niraparib 200 mg + Cetrelimab 480 mg (N=6) | Combination 1: Part 2 (Dose Expansion): Cohort 1A: BM+: Niraparib 200 mg + Cetrelimab 480 mg (N=21) | Combination 1: Part 2 (Dose Expansion): Cohort 1B: BM-: Niraparib 200 mg + Cetrelimab 480 mg (N=11) | Combination 2: Cohort 2A: Niraparib+Abiraterone Acetate+Prednisone (N=8) | Combination 2: Cohort 2C: Niraparib+Abiraterone Acetate+Prednisone (N=9) | Combination 2: Cohort 2D: Niraparib+Abiraterone Acetate+Prednisone (N=6) | Combination 2: Cohort 2C: HRR Negative: Niraparib + Abiraterone Acetate + Prednisone (N=1) | Combination 3: Cohort 1A: Niraparib + Abiraterone Acetate, SA (N=17) | Combination 3: Cohort 1B: Niraparib + Abiraterone Acetate, FDC1-RS (G010) (N=17) | Combination 3: Cohort 2: Niraparib + Abiraterone Acetate, FDC2-RS (G012) (N=17) | Combination 3: Cohort 3: Niraparib + Abiraterone Acetate, FDC1-LS (N=17)
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 7 | 4 | 4 | 6 | 2 | 1 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 5 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 5 | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 5 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 6 | 3 | 5 | 6 | 0 | 0 | 1 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye Pain (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye Swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular Hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 2 | 13 | 3 | 3 | 6 | 3 | 1 | 2 | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 1 | 1 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Angiodysplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gingival Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hiatus Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip Dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 9 | 1 | 3 | 4 | 2 | 0 | 2 | 2 | 1 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tongue Coated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 8 | 2 | 4 | 3 | 0 | 1 | 0 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 2 | 1 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 1
Chest Discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 3 | 10 | 8 | 3 | 5 | 4 | 1 | 2 | 0 | 3 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection Site Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 4 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Swelling (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Temperature Intolerance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Candida Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Tooth Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 2 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation Proctitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alpha 1 Globulin Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alpha 2 Globulin Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 3 | 4 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 1 | 6 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Chloride Decreased (Investigations) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Corticotrophin Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Corticotrophin Increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 1 | 4 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Thyroid Stimulating Hormone Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Urea Increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cortisol Decreased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibrin D Dimer Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lipase Increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroxine Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroxine Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tri-Iodothyronine Decreased (Investigations) | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin T Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 10 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Abnormal Loss of Weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 4 | 13 | 7 | 1 | 4 | 2 | 1 | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 6 | 3 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 2
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 2 | 5 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Facial Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 3 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental Impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Taste Disorder (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 5 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mood Altered (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Micturition Urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urine Flow Decreased (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic Discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Testicular Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 4 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 4 | 3 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT03431350/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT03431350/SAP_002.pdf